CLINICAL TRIAL: NCT02651688
Title: A Randomized, Double Blind, Placebo-Controlled, Multi-Center Study in Men With Acquired Hypogonadotropic Hypogonadism to Compare Changes in Body Composition and Metabolic Parameters With Diet and Exercise in Conjunction With Treatment With 12.5 mg or 25 mg Enclomiphene
Brief Title: A Multi-Center Study in Men With Acquired Hypogonadotropic Hypogonadism to Compare Changes in Body Composition and Metabolic Parameters With Diet and Exercise in Conjunction With Treatment With 12.5 mg or 25 mg Enclomiphene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZA-205
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Acquired Hypogonadotropic Hypogonadism; Obesity
MeSH Terms: conditions — Obesity | interventions — Enclomiphene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enclomiphene 12.5 mg (Experimental): Enclomiphene 12.5 milligram (mg) capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participant followed a commercial diet plan and exercised with a personal trainer at least 3 times a week.
  Interventions: Drug: Enclomiphene
- Enclomiphene 25 mg (Experimental): Enclomiphene 25 mg capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participant followed a commercial diet plan and exercised with a personal trainer at least 3 times a week.
  Interventions: Drug: Enclomiphene
- Placebo (Placebo Comparator): One matching placebo capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participant followed a commercial diet plan and exercised with a personal trainer at least 3 times a week.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — One matching placebo capsule daily in the morning with approximately 8 ounces of water for up to 12 months.
  Arms: Placebo
Drug: Enclomiphene — Enclomiphene capsule daily in the morning with approximately 8 ounces of water for up to 12 months.
  Arms: Enclomiphene 12.5 mg; Enclomiphene 25 mg

SUMMARY:
The purpose of this study is to compare the effects of 12 months of treatment with enclomiphene 12.5 mg, 25 mg, or placebo capsules on body composition and metabolic parameters in overweight men with acquired hypogonadotropic hypogonadism [confirmed morning testosterone (T) ≤300 ng/dL] following a 6 month diet and 15 month exercise program.

DETAILED DESCRIPTION:
To compare the effects of 12 months of treatment with enclomiphene 12.5 mg, 25 mg, or placebo capsules on body composition and metabolic parameters in overweight men with acquired hypogonadotropic hypogonadism (confirmed morning T≤300 ng/dL) following a 6 month diet and 15 month exercise program. Participants must not have been treated with testosterone products in the 6 months prior to the study and must not ever have used testosterone products for a year or longer.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (Body Mass Index (BMI) 30 to 42 (kg/m^2) inclusive) males age 18 to 60 inclusive.
* Waist circumference ≥ 40 inches (101.6 cm).
* Previously or concurrently diagnosed as having secondary hypogonadism.
* Must have 2 morning testosterone assessments at Visit 1, collected before 10 AM, 2-4 days apart, and both of which must be ≤ 300 (ng/dL).
* Luteinizing hormone (LH) >1.4 and < 9.4 milli International units per milliliter (mIU/mL) (at Visit 1 only).
* Glycated hemoglobin A1c (HbA1c) ≤7.5.
* Stable weight for last 3 months (+/- 10 pounds).
* Participant lives or works within 10 miles of the gym that will be used for the study.
* Must be fit enough to participate in the fitness program.
* Ability to complete the study in compliance with the protocol requirements.
* Ability to understand and provide written informed consent.

Exclusion Criteria:

* Any use of testosterone products (injectable, pelleted, transdermal or sublingual) in the 6 months prior to the study or any prior use of testosterone products for 12 months or longer at any time.
* Use of testosterone, Clomid, 5α-reductase inhibitors, human chorionic gonadotropin (hCG), androgen, estrogen, anabolic steroid, dehydroepiandrosterone (DHEA), or herbal hormone products during the study.
* Use of Clomid in the past year.
* Known hypersensitivity to Clomid.
* Allergy to soy, peanuts or latex.
* Chronic use of glucocorticoids (chronic use of inhaled or topical glucocorticoids is acceptable).
* History of drug abuse or chronic narcotic use including methadone.
* A recent history of alcoholism or illegal substance or steroid abuse (<2 years) or presence of moderate alcohol use (>21 drinks per week).
* Use of an investigational drug or product, or participation in a drug or medical device research study within 30 days prior to receiving study medication.
* A hematocrit >54%.
* Presence or known history of hyperprolactinemia with or without a tumor (prolactin >20 ng/mL).
* Current or history of prostate cancer or a suspicion of prostate disease unless ruled out by prostate biopsy, or a prostate specific antigen (PSA)>3.6.
* Current or history of breast cancer.
* Uncontrolled hypertension based on the Investigator's assessment at screening.
* History of bulimia nervosa or binge eating.
* Participant has (had) a lap band or undergone gastric bypass surgery.
* Participant has celiac disease or gluten intolerance.
* Participant has Type I diabetes.
* Participant has any condition which in the opinion of the investigator would interfere with the participant's ability to provide informed consent, comply with study instructions, possibly confound interpretation of study results, or endanger the participant if he took part in the study.
* Enrolled and randomized (if applicable) in a previous enclomiphene study.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Chan, Study Director — Allergan
Locations (5):
- United States (5):
  - Albany, New York
  - Garden City, New York
  - Providence, Rhode Island
  - Riverton, Utah
  - Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Enclomiphene 12.5 mg: Enclomiphene 12.5 milligram (mg) capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participants followed a commercial diet plan and exercise with a personal trainer at least 3 times a week.
- Enclomiphene 25 mg: Enclomiphene 25 mg capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participants followed a commercial diet plan and exercise with a personal trainer at least 3 times a week.
- Placebo: One matching placebo capsule daily in the morning with approximately 8 ounces of water for up to 12 months. Participants followed a commercial diet plan and exercise with a personal trainer at least 3 times a week.
Period: Overall Study
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Started | 18 | 17 | 15
Completed | 16 | 12 | 12
Not Completed | 2 | 5 | 3
Not completed — Non-compliance | 0 | 0 | 1
Not completed — Principal Investigator (PI) decision | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one treatment (with either enclomiphene or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 15 | 50
Age, Continuous [Mean (Full Range); unit: years] — Population: Safety population included all participants who received at least one treatment (with either enclomiphene or placebo).
  years | 42.2 [26 to 61] | 44.9 [18 to 59] | 44.9 [28 to 54] | 44.0 [18 to 61]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Safety population included all participants who received at least one treatment (with either enclomiphene or placebo).
  Participants
    Male | 18 | 17 | 15 | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lean Body Mass (LBM) at Week 48
Description: LBM was assessed using dual-energy X-ray absorptiometry (DXA). A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: Intent to treat (ITT) population consisted of all participants randomized to treatment with enclomiphene or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
kg
  Baseline | 65.23 (7.08) | 65.60 (7.88) | 68.12 (7.43)
  Change from Baseline to week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to week 48 | 3.14 (4.03) | 2.40 (3.54) | 1.05 (4.10)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.7103, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.4529, Wilcoxon rank-sum test

2. Primary Outcome: Change From Baseline in Body Strength (Chest Press Weight) at Week 48
Description: Body strength was assessed from maximum chest and leg press weight achieved, using an inclined plane leg press and vertical chest press. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: ITT population consisted of all participants randomized to treatment with enclomiphene or placebo. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pounds (lbs)
  Baseline: number analyzed (Participants) | 17 | 14 | 14
  Baseline | 169.00 (56.46) | 180.93 (95.43) | 151.50 (63.68)
  Change from Baseline to Week 48: number analyzed (Participants) | 13 | 10 | 11
  Change from Baseline to Week 48 | 75.00 (28.80) | 76.90 (51.55) | 87.27 (50.61)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.9302, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.7509, Wilcoxon rank-sum test

3. Primary Outcome: Change From Baseline in Body Strength (Leg Press Weight) at Week 48
Description: as for outcome 2
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pounds (lbs)
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pounds (lbs)
  Baseline: number analyzed (Participants) | 17 | 15 | 14
  Baseline | 466.06 (291.7) | 464.20 (288.2) | 580.86 (264.2)
  Change from Baseline to Week 48: number analyzed (Participants) | 12 | 10 | 10
  Change from Baseline to Week 48 | 406.92 (222.2) | 323.80 (200.3) | 351.50 (216.2)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.5095, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.6230, Wilcoxon rank-sum test

4. Primary Outcome: Change From Baseline in Blood Luteinizing Hormone (LH) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the hormone parameter LH measured in milli-International Units per milliliter (mIU/mL). A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
mIU/mL
  Baseline | 3.93 (1.82) | 3.41 (0.93) | 3.51 (1.31)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | 2.40 (3.39) | 3.01 (4.70) | 0.83 (1.25)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.2960, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.2723, Wilcoxon rank-sum test

5. Primary Outcome: Change From Baseline in Blood Testosterone (T) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the hormone parameter T. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
ng/dL
  Baseline | 243.56 (55.03) | 218.24 (43.39) | 223.53 (58.01)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | 173.81 (130.7) | 237.17 (181.4) | 43.33 (59.50)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0034, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.0027, Wilcoxon rank-sum test

6. Primary Outcome: Change From Baseline in Blood Dihydrotestosterone (DHT) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the hormone parameter DHT. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram per deciliter (ng/dL)
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
nanogram per deciliter (ng/dL)
  Baseline | 18.78 (7.74) | 16.06 (5.76) | 15.73 (5.92)
  Change from Baseline to Week 48: number analyzed (Participants) | 15 | 12 | 12
  Change from Baseline to Week 48 | 15.13 (12.92) | 20.75 (15.21) | 4.25 (5.96)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0146, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.0018, Wilcoxon rank-sum test

7. Primary Outcome: Change From Baseline in Blood Estradiol (E2) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the hormone parameter E2. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pg/mL
  Baseline | 50.04 (16.80) | 48.43 (15.15) | 45.49 (12.05)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 11
  Change from Baseline to Week 48 | -3.00 (28.02) | 13.03 (26.20) | -11.46 (15.41)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.1524, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.0227, Wilcoxon rank-sum test

8. Primary Outcome: Change From Baseline in Ratio of Testosterone: Estradiol (T:E2) at Week 48
Description: The T:E2 ratio was calculated as the value of T/value of E2 using the same units. A positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
ratio
  Baseline | 5.26 (1.73) | 4.93 (1.96) | 5.21 (1.88)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 11
  Change from Baseline to Week 48 | 5.11 (7.57) | 2.89 (3.09) | 2.85 (3.36)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.5873, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.9509, Wilcoxon rank-sum test

9. Primary Outcome: Change From Baseline in Ratio of Dihydrotestosterone: Testosterone (DHT:T) at Week 48
Description: The DHT:T ratio was calculated as the value of DHT/value of T using the same units. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
ratio
  Baseline: number analyzed (Participants) | 18 | 17 | 14
  Baseline | 0.08 (0.02) | 0.08 (0.03) | 0.07 (0.03)
  Change from Baseline to Week 48: number analyzed (Participants) | 13 | 10 | 11
  Change from Baseline to Week 48 | 0.01 (0.03) | 0.00 (0.02) | 0.00 (0.02)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.4341, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 1.0000, Wilcoxon rank-sum test

10. Primary Outcome: Change From Baseline in Glycated Hemoglobin A1c (HbA1c) at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter HbA1c. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
percentage of HbA1c
  Baseline | 5.56 (0.35) | 5.95 (0.74) | 5.77 (0.32)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | -0.34 (0.37) | -0.54 (0.27) | -0.65 (0.28)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0220, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.3677, Wilcoxon rank-sum test

11. Primary Outcome: Change From Baseline in Blood Glucose Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter Glucose. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pg/mL
  Baseline | 98.39 (14.71) | 101.41 (10.69) | 97.93 (13.22)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | -1.81 (16.69) | -5.25 (8.70) | -4.33 (13.29)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.9074, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.4517, Wilcoxon rank-sum test

12. Primary Outcome: Change From Baseline in Blood C-reactive Protein (CRP) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter CRP. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
mg/dL
  Baseline | 0.25 (0.22) | 0.35 (0.41) | 0.35 (0.35)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | 0.06 (0.50) | -0.05 (0.29) | -0.15 (0.25)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.2962, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.3261, Wilcoxon rank-sum test

13. Primary Outcome: Change From Baseline in Blood Interleukin-6 (IL-6) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter IL-6. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pg/mL
  Baseline: number analyzed (Participants) | 17 | 15 | 14
  Baseline | 2.23 (0.98) | 3.38 (1.76) | 2.75 (1.25)
  Change from Baseline to Week 48: number analyzed (Participants) | 13 | 7 | 9
  Change from Baseline to Week 48 | 0.56 (1.55) | -0.21 (1.50) | -0.78 (1.57)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0450, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.2235, Wilcoxon rank-sum test

14. Primary Outcome: Change From Baseline in Blood Tumor Necrosis Factor Alpha (TNF-α) Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter TNF-α . A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
pg/mL
  Baseline | 1.77 (0.68) | 1.93 (1.19) | 1.94 (0.84)
  Change from Baseline to Week 48: number analyzed (Participants) | 15 | 12 | 12
  Change from Baseline to Week 48 | -0.63 (0.69) | -0.35 (0.88) | -0.70 (0.65)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.8260, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.4183, Wilcoxon rank-sum test

15. Primary Outcome: Change From Baseline in Blood Leptin Level at Week 48
Description: A blood sample was collected at Baseline and Week 48 for the assessment of the metabolic parameter leptin. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
ng/mL
  Baseline | 9.88 (4.64) | 16.55 (9.14) | 15.16 (4.65)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | 1.14 (5.81) | 2.63 (12.10) | -2.27 (11.27)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.1144, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.3263, Wilcoxon rank-sum test

16. Primary Outcome: Change From Baseline in Homeostatic Model of Assessment - Insulin Resistance (HOMA-IR) at Week 48
Description: The HOMA-IR is the product of the blood Glucose and Insulin levels, divided by a constant. HOMA-IR is expressed as the following: HOMA-IR = fasting serum insulin (μU/mL) × fasting plasma glucose (mmol/L)/22.5. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
units on a scale
  Baseline: number analyzed (Participants) | 16 | 12 | 15
  Baseline | 4.88 (3.59) | 4.99 (2.92) | 4.74 (2.16)
  Change from Baseline to Week 48: number analyzed (Participants) | 14 | 10 | 11
  Change from Baseline to Week 48 | -1.14 (4.50) | -0.75 (3.17) | -1.80 (2.01)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.1546, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.5732, Wilcoxon rank-sum test

17. Primary Outcome: Change From Baseline in Blood Quantose-Insulin Resistance (IR) Score at Week 48
Description: Quantose-IR is a laboratory-developed test that assesses insulin resistance. Quantose-IR score is based on a linear regression algorithm utilizing the quantitative measures (natural log transformed) of alpha-hydroxybutyrate, oleate, linoleoylglycerophosphocholine and insulin and was designed to estimate the natural log of insulin-induced glucose infusion rate normalized by whole body mass. The algorithm score is converted to the Quantose-IR score within a range of 1-120 by an arithmetic calculation where higher scores denote greater insulin resistance. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Quantose-IR score
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
Quantose-IR score
  Baseline: number analyzed (Participants) | 16 | 12 | 15
  Baseline | 75.74 (11.98) | 76.50 (8.40) | 78.05 (12.41)
  Change from Baseline to Week 48: number analyzed (Participants) | 15 | 12 | 12
  Change from Baseline to Week 48 | -3.96 (10.65) | -6.59 (17.41) | -6.50 (13.71)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.5581, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.5833, Wilcoxon rank-sum test

18. Primary Outcome: Change From Baseline in Body Mass Index (BMI) at Week 48
Description: BMI is calculated as weight (kg)/height(cm^2). A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
kg/cm^2
  Baseline | 35.45 (3.01) | 37.38 (3.62) | 38.05 (2.63)
  Change from Baseline to Week 48: number analyzed (Participants) | 15 | 11 | 12
  Change from Baseline to Week 48 | -1.43 (3.27) | -2.29 (2.78) | -4.38 (2.94)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0168, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.0364, Wilcoxon rank-sum test

19. Primary Outcome: Change From Baseline in Waist Circumference at Week 48
Description: A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
cm
  Baseline | 115.34 (7.12) | 120.87 (10.89) | 123.96 (12.09)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | -6.71 (6.68) | -6.52 (13.04) | -12.62 (10.59)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0992, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.1333, Wilcoxon rank-sum

20. Primary Outcome: Change From Baseline in Weight at Week 48
Description: A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 0) to Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
Number analyzed (Participants) | 18 | 17 | 15
kg
  Baseline | 114.13 (11.31) | 121.75 (13.76) | 124.58 (10.96)
  Change from Baseline to Week 48: number analyzed (Participants) | 16 | 12 | 12
  Change from Baseline to Week 48 | -4.36 (9.95) | -6.15 (9.46) | -14.51 (10.34)
Statistical Analysis 1: Comparison: Enclomiphene 12.5 mg vs Placebo; Test type: Superiority; p = 0.0139, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Enclomiphene 25 mg vs Placebo; Test type: Superiority; p = 0.0225, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: From the first dose of the study drug through 30 days of the treatment end date (approximately 13 months)
Arm/Group | Enclomiphene 12.5 mg | Enclomiphene 25 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/18 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 13/18 | 7/17 | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enclomiphene 12.5 mg (N=18) | Enclomiphene 25 mg (N=17) | Placebo (N=15)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Ischaemic stroke (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enclomiphene 12.5 mg (N=18) | Enclomiphene 25 mg (N=17) | Placebo (N=15)
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Night sweats (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 1
Coxsackie viral infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 2
Influenza (Infections and infestations) | 1 | 1 | 0
Viral pharyngitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Food poisoning (Infections and infestations) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0
Haematocrit increased (Investigations) | 1 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Laceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vasectomy (Surgical and medical procedures) | 0 | 0 | 1
Haemorrhoids (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2016-07-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02651688/SAP_000.pdf
  • Study Protocol (2016-12-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT02651688/Prot_001.pdf